CLINICAL TRIAL: NCT03275376
Title: Statin Combination Therapy in Patients Receiving Sorafenib for Advanced Hepatocellular Carcinoma: A Randomized Controlled Study
Brief Title: Statin Combination Therapy in Patients Receiving Sorafenib for Advanced Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow in patient enrollment
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Teng-Yu Lee, MD, PhD, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF16263B
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Overall Survival; Tumor Responses
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Statin treated group (Experimental)
  Interventions: Drug: Atorvastatin 10mg
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Atorvastatin 10mg — Atorvastatin or placebo will be administered according to randomized allocations.
  Arms: Statin treated group
Drug: Placebo Oral Tablet — Atorvastatin or placebo will be administered according to randomized allocations.
  Arms: Control group

SUMMARY:
Target therapy with sorafenib is the standard of treatment for advanced Hepatocellular carcinoma (HCC), but the patient survival time is still unsatisfactory. The aims of this study are to prove statins improve the tumor responses and overall survival for patients who receive sorafenib therapy for advanced HCC by a prospective randomized controlled study.

DETAILED DESCRIPTION:
Background:

Hepatocellular carcinoma (HCC) is the second leading cause of cancer death worldwide, including the condition in Taiwan, and the management of HCC is an important challenge in public health. Target therapy with sorafenib is the standard of treatment for advanced HCC (vascular invasion or extrahepatic metastasis), but the patient survival time is still unsatisfactory. In recent years, growing evidences, including mechanism analysis, have suggested the anitneoplastic effects of statin, and a recent pooled analysis found that statin use may be associated with improved survival in patients with metastatic rencal cell carcinoma. However, a prospective clinical trial of statin sorafenib combination therapy in the treatment of advanced HCC is lacking.

Aims:

1. To prove statins improve the overall survival for patients who receive sorafenib therapy for advanced HCC by a prospective randomized controlled study.
2. To prove statin can improve tumor responses and the progression free survival for patients who receive sorafenib therapy for advanced HCC by a prospective randomized controlled study.

Methods:

This randomized placebo-controlled study will prospectively enroll patients who receiving sorafenib therapy for advanced HCC in the Taichung Veterans General Hospital, and statin or placebo will be statin or placebo will be administered according to randomized allocations. Tumor responses, time to tumor progression, and survival time will be followed and recorded

ELIGIBILITY:
Inclusion Criteria:

1. Patients more than 40 years old
2. HCCs diagnosed by AASLD image criteria or pathology
3. HCCs in BCLC advanced stage, with portal vein thrombosis (VP3 or VP4) or extrahepatic metastasis
4. Not suitable or failed to locoreginal treatments for HCC
5. Child-Pugh score = or < 6
6. ECOG performance status (PST) 0-2
7. Serum bilirubin < 2 mg/dL and prothrombin time (PT) prolongation < 3 seconds
8. Will receive sorafenib therapy
9. Life expectancy > 3 months
10. Will follow the pregnancy prevention protocol

Exclusion Criteria:

1. HCC is considered for curative therapy
2. HCC with brain metastasis
3. History of systemic therapy for HCC
4. Indications for statin use, such as hyperlipidemia in cardiovascular diseases
5. Any local treatment for HCC within 4 weeks
6. Any active gastrointestinal bleeding within 4 weeks
7. Liver transplant history or concomitant immunosuppressive therapy
8. Concurrent any other malignancy
9. Allergy to sorafenib or statins
10. Pregnancy or lactation
11. Serum AST or ALT > 5x upper limit of normal
12. Known HIV infection
13. eGFR < 30 ml/min
14. Abnormal medical conditions that are unsuitable for study, such as uncontrolled hypertension, coronary arterial disease, or arrhythmia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
Overall survival | Three year

SECONDARY OUTCOMES:
Best tumor response | Three year
Progression free survival | Three year

CONTACTS AND LOCATIONS:
Overall Officials: Teng-Yu Lee, MD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Llovet JM, Ricci S, Mazzaferro V, et al. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med 2008;359:378-390. 2. Cheng AL, Kang YK, Chen Z, et al. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol 2009;10:25-34. 3. Cainap C, Qin S, Huang WT, et al. Linifanib versus Sorafenib in patients with advanced hepatocellular carcinoma: results of a randomized phase III trial. J Clin Oncol 2015;33:172-179. 4. Llovet JM, Decaens T, Raoul JL, et al. Brivanib in patients with advanced hepatocellular carcinoma who were intolerant to sorafenib or for whom sorafenib failed: results from the randomized phase III BRISK-PS study. J Clin Oncol 2013;31:3509-3516. 5. Singh S, Singh PP, Roberts LR, et al. Chemopreventive strategies in hepatocellular carcinoma. Nat Rev Gastroenterol Hepatol 2014;11:45-54. 6. Demierre MF, Higgins PD, Gruber SB, et al. Statins and cancer prevention. Nat Rev Cancer 2005;5:930-942. 7. Wu J, Wong WW, Khosravi F, et al. Blocking the Raf/MEK/ERK pathway sensitizes acute myelogenous leukemia cells to lovastatin-induced apoptosis. Cancer Res 2004;64:6461-6468. 8. Rao S, Porter DC, Chen X, et al. Lovastatin-mediated G1 arrest is through inhibition of the proteasome, independent of hydroxymethyl glutaryl-CoA reductase. Proc Natl Acad Sci U S A 1999;96:7797-7802. 9. El-Serag HB, Johnson ML, Hachem C, et al. Statins are associated with a reduced risk of hepatocellular carcinoma in a large cohort of patients with diabetes. Gastroenterology 2009;136:1601-1608. 10. Tsan YT, Lee CH, Wang JD, et al. Statins and the risk of hepatocellular carcinoma in patients with hepatitis B virus infection. J Clin Oncol 2012;30:623-630. 11. Chiu HF, Ho SC, Chen CC, et al. Statin use and the risk of liver cancer: a population-based case-control study. Am J Gastroenterol 2011;106:894-898.